CLINICAL TRIAL: NCT00593177
Title: A Multi-Center Randomized, Double-Blind, Placebo-Controlled Study of 0.10% or 0.05% PTH (1-34) Gel Versus Placebo Gel in the Treatment of Mild to Moderate Plaque Psoriasis.
Brief Title: A Safety and Efficacy Study of a Topical Gel for the Treatment of Mild to Moderate Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manhattan Pharmaceuticals (Industry)
Collaborators: Therapeutics, Inc. (Industry)
Responsible Party: Tatjana Lukic, M.D., M. Sc., Study Director, Manhattan Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAN-PTH (1-34)-USA-002; 095-3351-201
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2008-08-19 (Estimated); Status verified 2008-07

CONDITIONS: Psoriasis Vulgaris
Keywords: Plaque psoriasis; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Group 1 (Experimental): 0.05% PTH (1-34) Gel
  Interventions: Drug: PTH (1-34) Gel / Placebo Gel
- Treatment Group 2 (Experimental): 0.10% PTH (1-34) Gel
  Interventions: Drug: PTH (1-34) Gel / Placebo Gel
- Treatment Group 3 (Placebo Comparator): Placebo (Vehicle) Gel
  Interventions: Drug: PTH (1-34) Gel / Placebo Gel

INTERVENTIONS:
Drug: PTH (1-34) Gel / Placebo Gel — Topical dosing of gel twice daily for eight weeks.

SUMMARY:
The primary objective of the study is to assess the tolerability and efficacy of a 0.10% or 0.05% PTH (1-34) parathyroid hormone peptide gel in the treatment of mild to moderate plaque psoriasis in comparison to treatment with the placebo gel alone.

DETAILED DESCRIPTION:
This pilot study aims to confirm the results of a previous proof of concept study performed by Dr. Michael Holick using a different dosage form. The secondary objective is to determine if there is a dose dependent difference or trend in response between the two concentrations of PTH (1-34) peptide gel.

Subjects will be randomized to receive one of three treatment groups on a 1:1:1 basis. The three treatment groups are:

* Treatment Group 1: 0.05% PTH (1-34) Gel
* Treatment Group 2: 0.10% PTH (1-34) Gel
* Treatment Group 3: Placebo Gel

ELIGIBILITY:
Inclusion Criteria:

* Mentally competent and has completed an appropriately administered informed consent.
* Male or non-pregnant female outpatient between the ages of 18 to 65 years.
* If subject is a woman of childbearing potential, she must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline, and agree to use an effective, non-prohibited form of birth control for the duration of the study (stabilized on hormonal contraceptives for at least two months (e.g. oral, implant, injection, NuvaRing, patch), IUD, condom and spermicidal or diaphragm and spermicidal, abstinence, etc.).
* Willing and able to apply the assigned study medication as directed, comply with study instructions and commit to all follow-up visits for the duration of the study.
* Clinical diagnosis of stable plaque psoriasis for at least 3 months.
* Plaque psoriasis with a minimum of 2% affected BSA (excluding palms, soles, face, scalp, groin, axillae or other intertriginous areas).
* Subject's disease is suitable to be managed topically for the duration of the trial.
* Subject has a Target Plaque that must have:

  * a minimum of 16 cm2 in area
  * an Overall Disease Severity Score of 2 or 3
  * an induration score of 2 or 3
* Willing and able to avoid prolonged exposure of the designated treatment lesions to ultraviolet radiation (natural and artificial) for the duration of the study.
* In good general health and free of any disease state or physical condition which might impair evaluation of plaque psoriasis or which, in the investigator's opinion, exposes the subject to an unacceptable risk by study participation.

Exclusion Criteria:

* Female who is lactating, or is planning to become pregnant during the study.
* Has spontaneously improving or rapidly deteriorating plaque psoriasis.- Has guttate, pustular, erythrodermic, inverse or other non-plaque forms of psoriasis.
* Has used any psoriasis vaccine or has participated in an investigational study of any psoriasis vaccine.
* Has used any systemic immunomodulatory therapy known to affect psoriasis that DOES typically decrease immune cell populations (e.g. alefacept) within the 36 weeks prior to start of treatment.- Subject has used any systemic immunomodulatory therapy known to affect psoriasis that DOES NOT typically decrease immune cell populations (e.g. efalizumab, etanercept, infliximab, adalimumab, and any investigational anti-TNF or anti-IL-12/23 agents) within 12 weeks prior to start of treatment.
* Has used any photo-therapy (including laser), photo-chemotherapy or systemic psoriasis therapy (e.g. systemic corticosteroids, methotrexate, retinoids or cyclosporine) within 4 weeks prior to start of treatment.
* Prolonged exposure to natural or artificial sources (e.g. UVB, UVA, etc.) of ultraviolet radiation within 4 weeks prior to the start of treatment or is intending to have such exposure during the study, thought by the investigator likely to modify the subject's psoriasis.
* Has used topical anti-psoriatic therapy (including topical retinoids, corticosteroids, vitamin D derivatives, topical immunomodulators, coal tar or salicylic acid preparations) on the areas to be treated within 2 weeks prior to start of treatment.
* Has used emollients/moisturizers on areas to be treated within 2 days prior to the start of treatment.
* Has used lithium or hydroxychloroquine within 4 weeks prior to start of treatment.
* Currently using a beta-blocking medication (e.g. propranolol) with a dose that has not been stabilized for at least 3 months prior to the start of treatment.
* Has recently been on medications for osteoporosis including but not limited to bisphosphonates, calcitonin, teriparatide, androgen or other anabolic steroid therapy, fluorides, vitamin D >50,000 IU/week, within the past 6 months.
* May be unreliable including subjects who engage in excessive alcohol intake or drug abuse.- Subject has, in the opinion of the investigator, any clinically significant abnormalities in the clinical laboratory tests (serum chemistries, hematology or urinalysis) conducted at screening.- Subject has a history of hypercalcemia (consistent with elevated serum calciums above 10.5 mg/dl), illnesses that affect bone or calcium metabolism or recent nephrolithiasis or urolithiasis (within the previous 2 years).
* Has a history of radiation therapy involving the skeleton.
* Has a history of sensitivity to any of the ingredients in the study medications.
* Currently enrolled in an investigational drug or device study.
* Has used an investigational drug or an investigational device treatment within 30 days prior to start of treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
All efficacy variables graded will be evaluated. Individual parameters of psoriasis include Erythema (0-4 scale); Scaling (0-4 scale); Induration (0-4 scale); Pruritus (0-3 scale); and Overall Disease Severity Score (0-4 scale). | Weeks 1 to 8

SECONDARY OUTCOMES:
As this is the early stage trial in psoriatic subjects using this novel topical therapy, no specific primary or secondary endpoints are designated. | Weeks 1 to 8

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Lukic, M.D., M.Sc., Study Chair — Manhattan Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Therapeutics Clinical Research, San Diego, California
  - Advanced Dermatology and Cosmetic Surgery, Ormond Beach, Florida
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Dermatology Research Center Inc., Salt Lake City, Utah

REFERENCES:
- [Background] Holick MF, Chimeh FN, Ray S. Topical PTH (1-34) is a novel, safe and effective treatment for psoriasis: a randomized self-controlled trial and an open trial. Br J Dermatol. 2003 Aug;149(2):370-6. doi: 10.1046/j.1365-2133.2003.05437.x. PMID 12932245
- See also: Abstract — http://www.ncbi.nlm.nih.gov/sites/entrez?Db=pubmed&Cmd=ShowDetailView&TermToSearch=12932245&ordinalpos=2&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_RVDocSum